CLINICAL TRIAL: NCT02590289
Title: An Open-Label, Single-Dose, 4-Way Crossover, Bioavailability Study to Evaluate the Pharmacokinetics, Pharmacodynamics, and Food Effect of BBI-5000 Capsules in Healthy Adult Subjects
Brief Title: A Pharmacokinetic Study to Evaluate BBI-5000 Capsules and Food Effect in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fresh Tracks Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BBI-5000-CL-103
Record Dates: First submitted 2015-10-20; First posted 2015-10-29 (Estimated); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- BBI-5000 Dose 1 (Experimental): Low dose of BBI-5000
  Interventions: Drug: BBI-5000
- BBI-5000 Dose 2 (Experimental): Middle dose of BBI-5000
  Interventions: Drug: BBI-5000
- BBI-5000 Dose 3 (Experimental): High dose of BBI-5000
  Interventions: Drug: BBI-5000
- BBI-5000 Dose 4 (Experimental): High dose of BBI-5000
  Interventions: Drug: BBI-5000

INTERVENTIONS:
Drug: BBI-5000 — BBI-5000 low dose, middle dose, or high doses

SUMMARY:
To assess the pharmacokinetics of 3 doses and the food effect of a single high dose of BBI-5000 capsules in healthy adult subjects.

DETAILED DESCRIPTION:
This is an open-label, randomized, 4-period, 4-way crossover, 4-sequence study to evaluate the pharmacokinetics (PK) and food effect of BBI-5000 capsules in healthy adult subjects.

Participating subjects will receive a single oral dose of BBI-5000 followed by a washout period of 7-14 days between doses. The treatment period will be followed by 5-10 day follow-up period.

PK and PD will be assessed by blood sampling through 72 hours postdose.

Safety will be assessed through collection of vital signs, adverse events, physical examination, ECGs and clinical laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker
* Medically healthy
* 32.0 >= BMI >= 18.5 kg/m^2
* Weight >= 50 kg for males
* Weight >= 45 kg for females
* For a female of childbearing potential: either be sexually inactive for 14 days prior to the first dose and throughout the study or be using an acceptable birth control method as dictated by the study
* Willing to comply with protocol and understands study procedures outlined in the ICF

Exclusion Criteria:

* Subject is mentally or legally incapacitated or has significant emotional problems
* History or presence of medical or psychiatric disease
* History of any illness that might confound the results of the study
* History or presence of alcoholism or drug abuse
* History or presence of hypersensitivity or idiosyncratic reaction the the study drug excipient
* History or presence of lactose intolerance
* Pregnant or lactating females
* Seated blood pressure less than 90/40 mmHg or greater than 140/90 mmHg
* Seated heart rate lower than 40 bpm or higher than 99 bpm
* Unable to refrain from or anticipates the use of any drug
* Diet incompatible with the on-study diet
* Donation of blood or significant blood loss within 56 days prior to the first study dose
* Participation in another clinical trial within 28 days prior to the first study dose

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations after single dosing of BBI-5000 for BBI-5000 and 3 metabolites | Week 4
Area Under Curve (AUC) for BBI-5000 and 3 metabolites | Week 4
Maximum Plasma Concentration (Cmax) for BBI-5000 and 3 metabolites | Week 4
Time of Occurrence of Cmax (Tmax) | Week 4
Clearance (CL/F) | Week 4
Terminal plasma elimination rate constant for BBI-5000 and the 3 metabolites | Week 4
BBI-5000 concentrations in plasma after dosing in fed and fasted conditions | Week 4
Half-life for BBI-5000 and the 3 metabolites | Week 4

SECONDARY OUTCOMES:
Safety and tolerability as measured by assessment of treatment-related adverse events, safety laboratory, vital signs, electrocardiogram and physical examination results | Week 4

OTHER OUTCOMES:
Eosinophil shape change in whole blood as measured by dose and exposure-related dependent changes over time | Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Hussey, PharmD, Study Director — Fresh Tracks Therapeutics, Inc.
Locations (1):
- Celerion Inc., Lincoln, Nebraska, United States